CLINICAL TRIAL: NCT05003544
Title: Comparıson Of PENG Block wıth Intra-articular And Quadratus Lumborum Block İn Primary Total Hip Arthroplasty: : Randomized Controlled Double Blinded Trial Trial
Brief Title: Comparıson Of PENG Block wıth Intra-articular And Quadratus Lumborum Block İn Primary Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-2021/14
Record Dates: First submitted 2021-08-03; First posted 2021-08-12 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-09

CONDITIONS: Hip Arthropathy
Keywords: PENG block; intra-artikuler; Quadrotus lumborum block; Hip Arthropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PENG BLOCK ( Group A) (Active Comparator): A regional block will be applied while the patient is in the supine position. A curvilinear low-frequency ultrasound probe (2-5MHz) will initially be placed in a transverse plane on the AIIS and then rotate the probe approximately 45 degrees counterclockwise to align with the pubic ramus. In this view, IPE, iliopsoas muscle and tendon, femoral artery and pectineus muscle will be observed. A 22 gauge, 80 mm needle will be inserted from lateral to medial in an in-plane approach to place the psoas tendon anteriorly and posteriorly in the musculofacial plane between the pubic ramus. Following negative aspiration, a local anesthetic solution (20ml bupivacaine 0.5%) will be injected.
  Interventions: Procedure: Group A
- Intra-articular( Group B) (Active Comparator): It will be applied to the intra-articular region by the surgeon at the end of the operation. A volume of 60 ml (30 ml of 0.5% bupivacaine and 30 ml of 0.9% NaCl)
  Interventions: Procedure: Group B
- Quadratus lumborum block ( Group C) (Active Comparator): The patient will be in the lateral position. A low-frequency convex probe will be vertically attached above the iliac crest and a needle will be inserted in-plane from the posterior edge of the convex probe through the quadratus lumborum in an anteromedial direction. The needle tip will be placed between the psoas major muscle and the quadratus lumborum muscle. After negative aspiration, 30 mL of 0.5 % of bupivacaine will be injected into the fascial plane incrementally, aspirating every 5 ml.
  Interventions: Procedure: Group C

INTERVENTIONS:
Procedure: Group A — PENG BLOCK
  Arms: PENG BLOCK ( Group A)
Procedure: Group B — Intra-articular
  Arms: Intra-articular( Group B)
Procedure: Group C — Quadratus lumborum block
  Arms: Quadratus lumborum block ( Group C)

SUMMARY:
90 patients ASA I-III, undergoing Total hip arthroplasty (THA) under spinal anesthesia, will be randomly assigned into one of three groups, namely group A (n=30), where an PENG block, group B (N:30) where an inra-articuler, and group C (n=30) where Quadratus lumborum block will be performed preoperatively. All patients will receive a standardized postoperative analgesia regimen. NRS scores will be evaluated in static and dynamic conditions during the first 48 hours postoperatively.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is the second most common joint replacement surgery, partly due to the aging population. The primary aim of this study is to compare the analgesic efficacy of Pericapsular nerve group (PENG) block with intra-articular and Quadrotus lumborum block (QLB). Regional anesthesia (RA), such as the recently described pericapsular nerve group (PENG) block, may provide additional analgesic benefit in this situation. Pericapsular nerve group (PENG) block is a new regional anesthesia technique to provide analgesia after hip fractures and hip arthroplasty. The aim of this single-center, double-blind, randomized controlled trial is to confirm the efficacy of PENG block for postoperative recovery after primary THA.

Routine multimodal analgesia will be used for postoperative analgesia

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA ) I-III

Exclusion Criteria:

* Previous operation on the same hip
* Hepatic or renal insufficiency
* Younger than 18 years old and older than 85
* Patients undergoing general anesthesia
* Allergy or intolerance to one of the study medications
* BMI >40
* ASA IV
* Chronic gabapentin/pregabalin use ( regular use for longer than 3 months)
* Chronic opioid use ( taking opioids for longer than 3 months, or daily oral morphine equivalent of >5 mg/day one month

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) scores | 48 Hours
  Range 0-10, 0=no pain, 10=the worse pain ever

SECONDARY OUTCOMES:
Opioid consumption | 3-6-8-12-24 and 48 hours
  Analgesic consumption
Static and dynamic pain | 3-6-8-12-24 and 48 hours
  Pain intensity at rest and during active movement using a numeric rating score (NRS) 0 = no pain and 10 = worst imaginable painranged from 0 to 10
Presence of quadriceps motor block (defined as paralysis or paresis ) | 3-6-12-24 hours after the block
  Quadriceps motor function will be tested with the patient supine and with the hip and knee flexed at 45º and 90º, respectively. The subject will be asked to extend the knee first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).
Hip adduction strength | 3-6-12-24 hours after the block
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1 and 2 points as decreases in strength of 0-20%, 21-70% and 71-90% compared to baseline measurement, respectively
Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depression | 3-6-12-24 hours after the block
  Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depressio
Patient satisfaction | 48 hours
  Patients asked whether they would choose the same anaesthetic management in a future operation: Yes/No
Quality of Recovery (QoR-40) score | measurements are obtained at 24 hours, 48 hours, and one week
  QoR-40, a 40-item questionnaire that provides a global score and sub-scores across five dimensions: patient support, comfort, emotions, physical independence, and pain. Each item is rated on a scale of 1-5, providing a minimum score of 40 and maximum of 200.
Mobilization time | 24 hour
  Mobilization time

CONTACTS AND LOCATIONS:
Locations (1):
- Tayfun Et, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikary SD, Short AJ, El-Boghdadly K, Abdelmalak MJ, Chin KJ. Transmuscular quadratus lumborum versus lumbar plexus block for total hip arthroplasty: A retrospective propensity score matched cohort study. J Anaesthesiol Clin Pharmacol. 2018 Jul-Sep;34(3):372-378. doi: 10.4103/joacp.JOACP_335_17. PMID 30386022